CLINICAL TRIAL: NCT06444126
Title: A Prospective Cohort Study Of The Incidence And Risk Factors Of Recurrent Febrile Seizures And Epilepsy Following Febrile Seizures
Brief Title: The Incidence And Risk Factors Of Recurrent Febrile Seizures And Epilepsy Following Febrile Seizures
Status: Recruiting | Type: Observational
Sponsor: Pham Ngoc Thach University of Medicine (Other)
Responsible Party: Principal Investigator, Bui Hieu Anh, Lecturer - Researcher, Pham Ngoc Thach University of Medicine
Other Study IDs: 16/23-BVNĐ2
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Febrile Seizures; Epilepsy in Children
MeSH Terms: conditions — Seizures, Febrile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Initial Febrile Seizures: The initial cohort included children hospitalized with their first febrile seizure

SUMMARY:
The goal of this observational study is to learn about the recurrence and development of epilepsy in children hospitalized with their first febrile seizures. The main questions it aims to answer are:

* What is the risk of recurrence after the first febrile seizure and what are the risk factors for recurrent febrile seizures in Vietnamese children?
* What is the risk of developing epilepsy later in life and what are the risk factors for developing epilepsy in Vietnamese children who have had febrile seizures?

DETAILED DESCRIPTION:
This was a single-center, longitudinal cohort study. Vietnamese children were prospectively identified for their first febrile seizures (FS) through the General Pediatric Department and Neurology Department of Children's Hospital 2 in Ho Chi Minh City between March and December 2023. This hospital is one of the largest tertiary pediatric hospitals in southern Vietnam with 1,400 beds, and receives about 90,000 admissions every year, with 800-1,000 cases of initial FS. After recruitment, the participants have been monitored for an average of two years to determine whether they experience recurring FS or develop epilepsy.

Sample size and sampling:

The sample size was calculated using a specific formula to estimate the incidence of FS recurrence in the cohort study. With the desired confidence level of 95%, an estimated error of 0.1, and an expected incidence of 31.8% based on a similar study conducted by Berg, the minimum sample size required was determined to be 385 participants. The sample size was also estimated based on the number of events per predictor in regression models, with at least 10 events per predictor recommended by Peduzzi et al. For the recurrent FS outcome, we have 12 potential predictor variables including age of onset, male gender, prematurity, low birth weight, neurodevelopmental abnormality, family history of FS or epilepsy, temperature, duration of fever at the time of the seizure, and characteristic of the first FS such as semiology, duration and number of seizures during the illness yielding approximately 120 cases to achieve the required sample size for estimating recurrence of FS. Besides that, we also have 16 potential predictor variables for the subsequent epilepsy outcome, including the above factors adding to the number of FS, and characteristics of all FS (first and recurrences). As such, we aimed to obtain at least 160 children. Finally, the overall sample size required at least 385 patients.

Convenience sampling was applied to recruit the participants. In detail, every weekday, the list of inpatient reports of the General Pediatric Department and Neurology Department on the electronic medical record database of Children's Hospital 2 was used to identify all children who had been diagnosed with FS and admitted to these departments. The investigator met with these children's parents or caregivers and asked a series of screening questions to confirm that they had not previously experienced febrile or unprovoked seizures. If the child had such a history, they were excluded from the study. The patients were then followed up until they recovered and were discharged from the hospital. At this point, the investigator made the final diagnosis of the first FS and assessed whether any exclusion criteria applied. If the patients were eligible for the study, the investigator obtained informed consent from their parents and proceeded to gather study data.

Data collection

The standardized questionnaire solicited child-related data including the age of onset, gender, perinatal history (i.e. age of gestation, birth weight, asphyxia, hospitalization at the neonatal intensive care unit), medical history (previous neurological diseases), family history of FS and epilepsy (including first relative and any relative); seizure-related data including semiology, duration, and number of seizures during the illness; and illness-related data including temperature, duration of fever at the time of the seizure, and the cause of fever. The interviewer obtained a comprehensive description of the seizure from either the parent or, if unavailable, from an eyewitness. Descriptions were compiled from both medical records and interviews, and additional clarification was sought, if necessary, by contacting the parent or witness again. Particular note was taken of the presence of asymmetrical features involving a unilateral arm, leg, or face (or some combination) or an eye deviation to one side, even if the fit later became bilateral tonic-clonic. Those seizures were classified as focal-onset seizures according to the ILAE classification in 2017. The presence of Todd's paresis (paralysis of one limb or one side of the body or a gaze palsy in the immediate postictal period) was considered indicative of a focal seizure. The study used medical records to gather information on seizures, associated symptoms, diagnosis, and temperature.

At the time of the first FS, a detailed neurologic examination and Denver II developmental screening test were conducted by a pediatrician. Test Denver II is a scale to assess the psychomotor development of children under 6 years old, which is validated and used in clinical practice in Vietnam. Test Denver II is a fairly comprehensive assessment of child development and focuses on 4 areas: personal-social, fine motor-adaptive, language, and gross motor. The interpretation of the test results indicates an obvious developmental delay if there are delayed items in at least two areas, with each area having a minimum of two items. A child is considered to have a suspected developmental delay if there are delayed items in one area with at least two items. If there are no signs of suspected or delayed development as described above, the child is considered normal. Developmental Quotient (DQ) is a calculation that reflects the rate of development in any given area and represents the percentage of normal development present at the time of testing.

Developmental Quotient (DQ)= (Developmental age (DA))/(Chronological age (CA)) x 100%

Lumbar puncture was performed only in cases that were indicative of meningitis or encephalitis, whereas neuroimaging (computerized tomography [CT] or magnetic resonance imaging [MRI]) was performed on children with focal seizures, febrile status epilepticus, or abnormal neurologic examination. Children who experience their first FS in our setting usually do not undergo an electroencephalography (EEG).

Following the initial interview, parents were contacted every three months to determine whether their child had experienced any further seizures and the circumstances under which they occurred. If a febrile seizure recurs or an afebrile seizure occurs, parents can report it immediately and directly to the investigator. Descriptions of the recurrent seizures were obtained in the same manner as for the initial FS. Whenever possible, we also obtained documentation of the recurrence from the medical record. Our goal was to follow children for an average of two years from the initial FS. We considered a seizure unprovoked if there were no acute precipitating circumstances to which the seizure could reasonably be attributed. According to the ILAE practical clinical definition from 2014, epilepsy is characterized by having two unprovoked seizures that are more than 24 hours apart. Children were censored from further analysis if they experienced an unprovoked seizure or were lost to follow-up.

Ethical considerations

The study protocol was approved by the Ethical Committee of Children's Hospital 2 (124/ GCN-BVNĐ2). and written consent was obtained from all participants. Informed consent was obtained from all study participants and their parents/caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Children had a diagnosis of first febrile seizure based on the definition of the International League Against Epilepsy (ILAE) in 1993. That was a seizure occurring in childhood after one month of age associated with a febrile illness not caused by an infection of the central nervous system, without previous neonatal seizures or a previous unprovoked seizure, and not meeting the criteria for other acute symptomatic seizures. Fever is clinically a temperature of at least 38°C by any method as recorded either in the emergency department, outpatient clinics, or as noted in the medical history, as well as measured upon admission to the inpatient departments.
* Patients were between 1 month and 8 years of age
* Agreement from parents with written informed consent

Exclusion Criteria:

* Febrile paroxysmal events were atypical for seizures
* Underlying neurological conditions that increase the likelihood of epilepsy
* Unwillingness to return for follow-up

Ages: 1 Month to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children, who had a diagnosis of first febrile seizure at discharge from the General Pediatric Department and Neurology Department of Children's Hospital 2
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
The incidence and risk factors of the recurrence of febrile seizures | 2 years
  Following the initial interview, parents were contacted every three months to determine whether their child had experienced any further seizures and the circumstances under which they occurred. If a febrile seizure recurs or an afebrile seizure occurs, parents can report it immediately and directly to the investigator.
The incidence and risk factors of the epilepsy following febrile seizures | 2 years
  We considered a seizure unprovoked if there were no acute precipitating circumstances to which the seizure could reasonably be attributed. According to the ILAE practical clinical definition from 2014, epilepsy is characterized by having two unprovoked seizures that are more than 24 hours apart

CONTACTS AND LOCATIONS:
Overall Officials: Hong Kim Tang, M.D, Ph.D, Study Director — Pham Ngoc Thach University of Medicine; Anh Hieu Bui, M.D, Principal Investigator — Pham Ngoc Thach University of Medicine; Van Khanh Le, M.D, Ph.D, Principal Investigator — Pham Ngoc Thach University of Medicine
Locations (1):
- Children's Hospital 2, Ho Chi Minh City, Vietnam